CLINICAL TRIAL: NCT06654856
Title: A Prospective, Multicenter, Single Group, Open-label and Observational Study to Evaluate the Effectiveness and Safety of Dong-A Opalmon® Tablet in Patients With Acquired Lumbar Spinal Stenosis
Brief Title: The Effectiveness and Safety of Dong-A Opalmon® Tablet in Patients With Acquired Lumbar Spinal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OMT_LSS_OS
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dong-A Opalmon® Tab

SUMMARY:
This study is to evaluate the Effectiveness and Safety of Dong-A Opalmon® Tablet in Patients With Acquired Lumbar Spinal Stenosis

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 19 years
* Subjects with acquired Lumbar Spinal Stenosis who show normal results in the Straight Leg Raising (SLR) test and exhibit intermittent claudication, requiring treatment with Dong-A Opalmon® tab
* Subjects who voluntarily consent to participate in this observational study

Exclusion Criteria:

* Subject for whom the medicinal products administration is contraindicated according to the approved domestic drug information: Pregnant women or those who may be pregnant, Subject with genetic disorders such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects considered as unsuitable for participation in this observational study by the principal investigator or sub-investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who require treatment of Dong-A Opalmon® tab due to acquired Lumbar Spinal Stenosis
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score of 'Symptom severity' and 'Physical function' items in Zurich Claudication Questionnaire at 8 weeks | Change from baseline at 8 weeks
  The total score for 'Symptom severity' is rated on a scale from 7 to 35 points, with higher score denoting more severe symptoms.
  The total score for 'Physical function' is rated on a scale from 5 to 20 points, with higher score denoting more severe disability.

SECONDARY OUTCOMES:
Mean score for 'Satisfaction' item in Zurich Claudication Questionnaire at 8 weeks | At 8 weeks
  The total score for 'Satisfaction' is rated on a scale from 6 to 24 points, with higher score denoting lower rate of satisfaction.
Change from baseline in Oswestry Disability Index score at 8 weeks | Change from baseline at 8 weeks
  The score for Oswestry Disability Index is rated on a scale from 0% to 100%, with higher score denoting more severe disability in everyday life.
Change from baseline in score for first question (how much can you walk) of Zurich Claudication Questionnaire Part 2 'Physical Function' at 8 weeks | Change from baseline at 8 weeks
  The score is rated on a scale from 1 to 4 points with higher score denoting more difficulty in walking.

CONTACTS AND LOCATIONS:
Locations (1):
- VHS Medical Center, Seoul, South Korea